CLINICAL TRIAL: NCT07270861
Title: A Multicenter, Non-interventional, Two-cohort Study to Describe Real-world Treatment Patterns and Outcomes in Patients With Peripheral T-cell Lymphoma
Brief Title: Real-world Outcomes of Peripheral T-cell Lymphoma: A Multicenter Retrospective and Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Rong Tao, Professor & Chief, Fudan University
Other Study IDs: SHCA-PTCL-202501
Record Dates: First submitted 2025-11-15; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Peripheral T-Cell Lymphoma
Keywords: T-cell lymphoma; Retrospective cohort; Prospective cohort; Epidemiology; Biomarkers
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Peripheral blood sample，tumor biopsy sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A (Retrospective): A retrospective cohort of cases diagnosed between 2010 and 2024, assembled from medical-record data.
  Target enrollment: 1,300-1,500 patients.
  Interventions: Other: Observational
- Cohort B (Prospective): A prospective cohort of patients newly diagnosed between 2025 and 2030, ensuring ≥5-year follow-up for all survivors.
  Target sample size: 1,000-1,500 cases, estimated from participating centers' annual diagnostic volumes over a 5-year accrual period. The cohort should be multidimensionally representative, including: (i) geographic coverage across North, East, South, Southwest, and Northeast China; (ii) hospital tiers with tertiary ("Class III Grade A") institutions as the core and selective inclusion of prefecture-level hospitals; and (iii) economic diversity spanning regions with differing levels of socioeconomic development.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
This study aims to characterize the epidemiology, clinicopathologic features, and survival outcomes of Chinese patients with PTCL; to develop and validate prognostic models to this population; to compare the real-world effectiveness and safety of alternative therapeutic strategies; to elucidate molecular mechanisms underlying treatment resistance and relapse; to identify actionable targets and predictive biomarkers.

DETAILED DESCRIPTION:
Due to disease heterogeneity and variability in clinical practice, establishing a large-scale Chinese PTCL database to characterize real-world treatment patterns and clinical outcomes is a critical undertaking. A retrospective cohort will define the clinical epidemiology of the disease, while a prospective cohort will delineate current treatment pathways and outcomes in routine practice and explore the molecular features of PTCL in the Chinese population, thereby providing evidence to support precision therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, with a histopathologic diagnosis of PTCL (any subtype per WHO 2016 classification of hematolymphoid neoplasms).
* Cohort A: Patients diagnosed and treated at participating centers between 2010 and 2024.
* Cohort B: Patients newly diagnosed from October 2025 onward.
* Availability of basic diagnostic and treatment records .

Exclusion Criteria:

* Indeterminate diagnosis or missing pathology report.
* Patients diagnosed at an outside institution who did not receive their primary treatment and follow-up at a participating center.
* Diagnoses of NK/T-cell lymphoma or primary cutaneous T-cell lymphomas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter, non-interventional, two-cohort study comprising a retrospective cohort (A) and a prospective cohort (B). We will include patients with a histopathologic diagnosis of peripheral T-cell lymphoma that meets the 2016 WHO criteria, excluding NK/T-cell lymphoma and primary cutaneous T-cell lymphomas. Eligible cases must have complete medical records and follow-up data.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Distribution of PTCL Histological Subtypes according to WHO 2016 Classification | Baseline (at the time of enrollment or diagnosis)
  The number and percentage of participants diagnosed with each specific subtype of Peripheral T-Cell Lymphoma (e.g., PTCL-NOS, AITL, ALCL, ENKTL, etc.). Diagnosis is confirmed by pathological review based on the WHO Classification of Tumours of Haematopoietic and Lymphoid Tissues (Revised 4th edition, 2017).
Overall Survival (OS) | 5 year after diagnosis
  OS is defined as the time from the date of pathological diagnosis to the date of death from any cause. For patients who are lost to follow-up, survival time will be censored at the date of last contact.
Progression-Free Survival (PFS) | 5 year after diagnosis
  PFS is defined as the time from the date of pathological diagnosis to the date of the first documented disease progression (PD) or death from any cause, whichever occurs first. Disease progression is assessed based on the investigator's evaluation of radiological and clinical data.

SECONDARY OUTCOMES:
Frequency of Specific Genetic Mutations | Up to 5 years (at Baseline and at time of Disease Progression/Relapse)
  Evaluation of the number and percentage of participants carrying specific genetic alterations. Key biomarkers to be assessed include:
  Gene Mutations: TET2, DNMT3A, IDH2, RHOA, TP53, EZH2, and genes related to the PI3K-AKT pathway, assessed by Next-Generation Sequencing (NGS) or ct-DNA analysis. Correlations between these biomarkers and clinical outcomes (response, survival) will be analyzed.
Expression levels of biomarker proteins | Up to 5 years (at Baseline and at time of Disease Progression/Relapse)
  Protein/Pathological Markers: Expression of PD-1/PD-L1, CD30, Ki-67 proliferation index, and EBV status, assessed by Immunohistochemistry (IHC) or In Situ Hybridization (ISH). Correlations between these biomarkers and clinical outcomes (response, survival) will be analyzed.
Incidence of Treatment-Emergent Adverse Events (TEAEs) assessed by CTCAE v5.0 | Up to 5 years
  Safety will be assessed by recording the number of participants with adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. This includes treatment-related deaths and incidence of second primary malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Result] Vose J, Armitage J, Weisenburger D; International T-Cell Lymphoma Project. International peripheral T-cell and natural killer/T-cell lymphoma study: pathology findings and clinical outcomes. J Clin Oncol. 2008 Sep 1;26(25):4124-30. doi: 10.1200/JCO.2008.16.4558. Epub 2008 Jul 14. PMID 18626005